CLINICAL TRIAL: NCT03254160
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled 42-Day Treatment Study to Evaluate the Effect of DNS-3379 on Upper Extremity Motor Function Following Ischemic Stroke
Brief Title: DNS-3379 vs. Placebo in Stroke Rehabilitation
Acronym: SPIRIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative
Sponsor: Dart NeuroScience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNS-3379-201
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Rehabilitation; Ischemic
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DNS-3379 (0.5mg) (Experimental)
  Interventions: Drug: DNS-3379
- DNS-3379 (2.5mg) (Experimental)
  Interventions: Drug: DNS-3379
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNS-3379 — DNS-3379
  Arms: DNS-3379 (0.5mg); DNS-3379 (2.5mg)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel group outpatient 42-day treatment study that will utilize standard stroke rehabilitation outcome measures to evaluate the effect of DNS-3379 on upper extremity motor recovery in subjects following ischemic stroke.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects who have experienced an ischemic stroke documented by CT or MRI resulting in upper extremity deficit that warrants the need for rehabilitation therapy.
* Medically stable subjects, with expected survival > 12 months, who are able to be randomized to study drug beginning between 1 and 52 weeks (i.e., 7 to 365 days) post-stroke.
* Mild to moderately severe upper extremity motor impairment.
* mRS score of 1 to 4 from index stroke.
* Mini Mental State Examination (MMSE) score of ≥ 22.

Main Exclusion Criteria:

* Residual motor deficit from any prior stroke
* Hemorrhagic stroke. Ischemic stroke with limited hemorrhagic conversion (i.e., petechial hemorrhage or micro-hemorrhage) is acceptable.
* Severe or total sensory loss
* Moderate to severe aphasia and/or severe language deficits
* Excessive spasticity in the affected elbow or change in oral spasticity treatment drugs within 2 weeks before the Screening Visit
* Prior botulinum toxin injection to any portion of the affected arm in the prior 3 months before the Screening Visit
* Major and active neurological, psychiatric, or medical diagnosis that is not adequately controlled and would likely reduce the safety of study participation or impact the subject's ability to comply with study protocol procedures in the opinion of the Investigator
* Any suicidal ideation during the subject's lifetime at any time prior to randomization including childhood (based on subject history), equivalent to type 2 on the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Received an investigational pharmacotherapy therapy within the past 3 months
* Heavy use of any tobacco-smoke emitting products (including but not limited to cigarettes, pipes, and cigars) within 30 days of Baseline.
* Pregnant or lactating females

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity Motor Function, Parts A-D | 42-days
Type and incidence of treatment emergent adverse events | 84-days
Safety Laboratory Assessments | 84-days
Vital signs and 12-lead ECG | 84-days

SECONDARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity Motor Function (Parts A-D) | 84-days
Nine-Hole Peg Test | 84-days
Action Research Arm Test | 84-days
Stroke Impact Scale | 84-days
Modified Rankin Scale | 84-days
Change in weight | 84-days
Columbia Suicide Severity Rating Scale | 84-days
Two-Minute Walk Test | 84-days
EQ-5D-5L | 84-days

OTHER OUTCOMES:
fMRI Imaging | 84-days

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (15):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Repatriation General Hospital, Daw Park, South Australia
  - Lyell McEwin, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincents Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Western Health, St Albans, Victoria
  - Albury/Wodonga Hospital, Wodonga, Victoria
  - Hollywood Hospital, Nedlands, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Auckland Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No